CLINICAL TRIAL: NCT04245033
Title: Evaluation of the Implementation and Effectiveness of Intermittent Preventive Treatment for Malaria Using Dihydroartemisinin-piperaquine on Reducing Malaria Burden in School Aged Children in Tanzania
Acronym: IPTsc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: National Malaria Control Program, Tanzania (Unknown)
Responsible Party: Principal Investigator, Dr. Geofrey Makenga, Research Scientist, National Institute for Medical Research, Tanzania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPTsc version 1
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: The study is an effectiveness-implementation hybrid trial to assess feasibility and effectiveness of IPTsc using DP against standard of care (control). Wards in the three study districts (Handeni DC, Handeni TC and Kilindi DC) will be the randomisation unit (clusters). Each ward will be randomised to implement IPTsc or not (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPTsc arm (Experimental): Dihydroartemisinin-Piperaquine (DP) for intermittent preventive treatment in school children (IPTsc) will be given in all wards in the IPTsc arm at an interval of four months, three times a year.
  Interventions: Drug: Dihydroartemisinin-Piperaquine (DP)
- Control (No Intervention): No intervention will be given to wards randomised in this arm

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine (DP) — Dihydroartemisinin-Piperaquine (DP) for intermittent preventive treatment of malaria in school children (IPTsc).
  Arms: IPTsc arm

SUMMARY:
In Tanzania, according to the National Malaria Control Programme (NMCP), malaria prevalence has declined from an average of 18.1% in 2008 to 7% in 2017, marked as an epidemiological transition from meso-endemic to hypo-endemic levels with variation across and within regions and/or councils. Children of school-age have become increasingly more vulnerable as compared to those aged less than five years. In high-transmission settings, up to 70% of school-aged children harbour malaria parasites which is mostly asymptomatic, accounting for around 50% of the mortality, 13-50% of all school absenteeism. The NMCP developed a supplementary malaria midterm strategic plan (SMMSP 2018-2020) to customise malaria interventions by stratifying the burden of malaria in Tanzania mainland and recommended use of Dihydroartemisinin-Piperaquine (DP) for intermittent preventive treatment in school children (IPTsc) in high malaria strata. The investigators plan to evaluate the implementation of IPTsc using DP, given three times a year, for evidence on the operational feasibility and effectiveness of IPTsc on clinical malaria incidence at a high endemic area in Handeni District Council (DC), Handeni Town Council (TC) and Kilindi DC of Tanga region, Tanzania.

The study is an effectiveness-implementation hybrid trial to assess feasibility and effectiveness of IPTsc using DP against standard of care (control). Wards in the three study districts (Handeni DC, Handeni TC and Kilindi DC) will be the randomisation unit (clusters). Each ward will be randomised to implement IPTsc or not (control). In all wards in the IPTsc arm, the interventional drugs (DP) will be given at an interval of four months, three times a year. For study evaluation of the impact of intervention, in each district representative randomly selected wards, will provide randomly selected school per ward (24 in total) to formulate part of evaluable children per intervention. Mixed design methods will be used to assess the feasibility and acceptability of implementing IPTsc as part of a more comprehensive school children health package.

The study is expected to be operationally feasible given existing school health programme for Neglected Tropical Disease (NTD) control and the school net programme (SNP). IPTsc is expected to increase malaria case management effectiveness and to have additional effect in reducing the burden of disease on top of optimal access to malaria case management (MCM) and malaria vector control (MVC) initiatives e.g. early diagnosis and treatment, and insecticide-treated nets (ITNs) coverage, respectively.

ELIGIBILITY:
The following eligibility criteria are used to enroll participants on for close monitoring follow ups assessing the effectiveness part of the study protocol.

Inclusion Criteria:

1. Includes parental/guardian informed consent
2. Assent by primary school children aged 11 years and above.
3. Aged 5-15 years.
4. Currently, lives within the pre-defined catchment area of study district; and
5. Will remain within the same area throughout the study period (preferably class five and below).

Exclusion Criteria:

1. Students at class 7
2. Currently enrolled in another study or participated in another investigational drug study within the last 30 days.
3. Known to have heart disease or a known cardiac ailment.
4. Reports known hypersensitivity to the study drugs.
5. Not willing to undergo all study procedures including physical examination and to provide blood samples as per this study protocol.
6. Having clinical features of severe anaemia
7. Febrile due to non-malaria illness at the time of recruitment.
8. Has apparent severe infection or any condition that requires hospitalization
9. Illness or conditions like hematologic, cardiac, renal, hepatic diseases which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study, including known G6PD deficiency and SS sickle cell.
10. Body weight < 12 kg

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4100 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Efficiency of school health teachers to deliver antimalarial drugs to school children in high endemic regions | 1 year from start of intervention
  Efficiency in terms of percentage of children given a complete dose in each round.
Clinical malaria incidence | from month 0 till month 12 of follow up
  Malaria incidence will be collected in terms of number of episodes a child gets malaria.

SECONDARY OUTCOMES:
Change in malaria incidence per 1000 population at local health facility level | from month 0 till month 12 of follow up
  Number of malaria episodes before and after intervention in a respective ward
Change from baseline in haemoglobin concentration | measured at month 12
  individual change in Haemoglobin before and after intervention
Number of participants with treatment-related adverse events | through study completion, an average of 1 year"
  Number of participants with treatment-related adverse events encountered by subjects per study arm
Cardio safety profile by QTc prolongation from baseline | Day 1, 2,3 and 7 after before and after dosing
  measured by ECG
Acceptability of IPTsc in communities with high malaria endemicities | At month 8 of implementation
  Through in depth interview in a guided questionnaire

OTHER OUTCOMES:
Proportion of school children with malnutrition | at month 0 (baseline) and at month 12.
  Weight and height will be combined to report BMI in kg/m^2, WHO's BMI z-score will be used to categorise nutrition status.

CONTACTS AND LOCATIONS:
Overall Officials: John P.A Lusingu, MD, PhD, Study Director — National Institute for Medical Research, Tanga, Tanzania; Ally Mohamed, MD, Study Director — National Malaria Control Programme, Tanzania; Geofrey Makenga, MD, Msc, PhD fellow, Principal Investigator — National Institute for Medical Research, Tanzania
Locations (1):
- Handeni Town Council, Handeni and Kilindi Districts, Tanga, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Makenga G, Mmbando B, Seth MD, Baraka V, Challe DP, Francis F, Mhina AD, Liheluka E, Minja DTR, Chiduo M, Mtove G, Mandara C, Gesase S, Segeja MD, Kamugisha M, Hayuma PM, Mbwana JR, Sebukoto H, Malabeja A, Tupa JB, Ngede SJ, Lusasi A, Chacky F, David A, Thawer SG, Mohamed A, Aaron S, Lazaro S, Molteni F, Nkayamba A, Bastiaens H, Van Geertruyden JP, Lusingu JPA. Implementation and effectiveness of intermittent preventive treatment in school aged children using dihydroartemisinin-piperaquine to reduce malaria burden: an implementation research of a cluster randomised trial in Tanzania. EClinicalMedicine. 2025 Nov 7;90:103628. doi: 10.1016/j.eclinm.2025.103628. eCollection 2025 Dec. PMID 41278241
- [Derived] Makenga G, Seth MD, Baraka V, Mmbando BP, Challe DP, Francis F, Mhina A, Minja DTR, Chiduo M, Mandara C, Liheluka E, Gesase S, Segeja M, Mtove G, Kamugisha M, Lusasi A, Chacky F, David A, Thawer S, Mohamed A, Lazaro S, Molteni F, Nkayamba A, Van Geertruyden JP, Lusingu JPA. Implementation research of a cluster randomized trial evaluating the implementation and effectiveness of intermittent preventive treatment for malaria using dihydroartemisinin-piperaquine on reducing malaria burden in school-aged children in Tanzania: methodology, challenges, and mitigation. Malar J. 2023 Jan 6;22(1):7. doi: 10.1186/s12936-022-04428-8. PMID 36609279